CLINICAL TRIAL: NCT00748813
Title: A Phase II, Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of Surface Antigen, Inactivated, Influenza Vaccine, Formulation 2008-2009, When Administered to Non-Elderly Adult and Elderly Sub
Brief Title: Safety and Immunogenicity of Surface Antigen, Inactivated, Influenza Vaccine Using the Strain Composition 2008/2009
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V71P7S; 2008-001079-31
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2011-12

CONDITIONS: Seasonal Influenza
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

ARMS (1):
- 1 (Other)
  Interventions: Biological: Influenza Vaccine, Formulation 2008-2009

INTERVENTIONS:
Biological: Influenza Vaccine, Formulation 2008-2009 — 1 dose of Surface Antigen, Inactivated, Influenza Vaccine, Formulation 2008-2009

SUMMARY:
Annual trial for registration influenza vaccine with the strain composition for season 2008/2009

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for enrollment into this study are male and female adults who are:

  1. ≥ 18 years of age, mentally competent, willing and able to give informed consent prior to study entry
  2. able to comply with all study requirements
  3. in good health as determined by:
* medical history
* physical examination
* clinical judgment of the investigator

Exclusion Criteria:

* They have any serious chronic or acute disease (in the judgment of the investigator) including but not limited to:

  1. Cancer, except for localized skin cancer;
  2. Advanced congestive heart failure;
  3. Chronic obstructive pulmonary disease (COPD);
  4. Autoimmune disease (including rheumatoid arthritis);
  5. Acute or progressive hepatic disease;
  6. Acute or progressive renal disease;
  7. Severe neurological or psychiatric disorder;
  8. Severe asthma.
* They have history of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine (e.g., to ovalbumin, chicken protein, chicken feathers, influenza viral protein, kanamycin and neomycin sulphate);
* They have a known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age) resulting, for example, from:
* receipt of immunosuppressive therapy (any parenteral or oral corticosteroid or cancer chemotherapy/radiotherapy) within the past 60 days and for the full length of the study;
* receipt of immunostimulants;
* receipt of parenteral immunoglobulin preparation, blood products and/or plasma derivates within the past 3 months and for the full length of the study;
* suspected or known HIV infection or HIV-related disease;
* They have a known or suspected history of drug or alcohol abuse;
* They have a bleeding diathesis or condition associated with prolonged bleeding time that in the investigator's opinion would interfere with the safety of the subject;
* Women who are pregnant, or women able to bear children but not willing to practice acceptable contraception for the duration of the trial (21 days);
* Within the past 12 months, they have:
* received more than one injection of influenza vaccine
* Within the past 6 months, they have:
* had laboratory confirmed influenza disease;
* received influenza vaccine;
* Within the past 4 weeks they have received:
* another vaccine;
* any investigational agent;
* They have any acute or chronic infection requiring systemic antibiotic treatment or antiviral therapy within the last 7 days; 1 - They have experienced an acute exacerbation of a COPD within the past 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of antibody response to each influenza vaccine antigen, as measured by Single Radial Hemolysis (SRH) test on Day 0 and on Day 21 | 21 days (-1/+5)

SECONDARY OUTCOMES:
Evaluation of safety | 21 days (-1/+5)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (3):
- Italy (3):
  - Site 1, Chieti
  - Site 2, Lanciano
  - Site 3, Pianiga